CLINICAL TRIAL: NCT03012958
Title: Utility of Lung Clearance Index Score as a Noninvasive Marker of Deployment Lung Disease
Acronym: LCI
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Cecile Rose Professor of Medicine, Principal Investigator, National Jewish Health
Other Study IDs: HS-2851
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Bronchiolitis; Pneumonitis; Dyspnea
MeSH Terms: conditions — Bronchiolitis; Pneumonia; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health control group: Who are 18 years or older, have no history of pre-existing lung disease, and report no respiratory illness in the four weeks preceding enrollment.
  This study consist of one visit: If the potential subject meets the Inclusion and exclusion then they will have the LCI testing.
  Interventions: Other: Lung clearance index (LCI)
- Deployment-related lung disease: Defined as the presence of unexplained chest symptoms in a deployer who, on surgical lung biopsy is found to have bronchiolitis or granulomatous pneumonitis without other known causes.
  This study consist of one visit: If the potential subject meets the Inclusion and exclusion then they will have the LCI testing.
  Interventions: Other: Lung clearance index (LCI)

INTERVENTIONS:
Other: Lung clearance index (LCI) — LCI is determined by the number of lung volume turnovers necessary to clear the lungs of an inert tracer gas such as nitrogen that is inhaled at the beginning of the test. The LCI is calculated by determining the cumulative expired volume (CEV) and then dividing the CEV by the functional residual capacity. Values of less than7.0 indicate normal values while an LCI greater than 7.0 is associated with heterogeneity in ventilation and distal airway abnormalities. The ability to detect peripheral airway disease may make LCI a better modality for detecting distal airways abnormalities seen on lung histopathology but often missed on traditional pulmonary function testing.

SUMMARY:
The purpose of this study is to learn more about new noninvasive ways of detecting lung disease in US Military personnel and people who worked as contractors during military operations in Iraq and Afghanistan. This study is looking at conducting a type of breathing test called the lung clearance index (LCI) test which is being investigated as a potential noninvasive way to detect the type of lung disease that may be seen in symptomatic deployers retuning from Iraq and Afghanistan.

DETAILED DESCRIPTION:
The healthy control group will comprise volunteers who are at least 18 years of age, have no history of pre-existing lung disease, and report no respiratory illness in the four weeks preceding enrollment.

The symptomatic deployers who have undergone lung biopsy and meet the case definition for deployment-related lung disease. A case of deployment-related lung disease is defined as the presence of unexplained chest symptoms in a deployer who, on a surgical lung biopsy, is found to have bronchiolitis or granulomatous pneumonitis without other known cause.

ELIGIBILITY:
Inclusion Criteria:

For the deployer group:

* presence of respiratory symptoms (cough, chest tightness, wheezing, shortness of breath or decreased exercise tolerance) following deployment
* history of deployment for Operation Iraqi Freedom, Operation Enduring Freedom or Operation New Dawn for greater than or equal to 6 weeks as either military personnel or a civilian contractor
* prior VATS biopsy-proven histologic abnormalities of small airways disease.

For the control group:

* no history of pre-existing lung disease
* no respiratory illness in the four weeks preceding enrollment

Exclusion Criteria:

For the deployer group:

* If on clinical evaluation they were found to have asthma, vocal cord dysfunction or other explanations for their respiratory symptoms and did not need to undergo surgical lung biopsy for diagnosis.
* unable to provide informed consent
* pregnant subjects

For the control group:

* pre-existing lung disease
* unable to provide informed consent
* pregnant subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic military deployers with deployment-related lung disease seen at National Jewish Health and healthy controls subjects.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
LCI parameters in symptomatic deployers compared to normal adults to determine whether LCI is an early marker of lung injury. | Up to 24 months
  Average of three acceptable trials

SECONDARY OUTCOMES:
Correlation between LCI score and the clinical characteristics of the population of deployers. | Up to 24 months
  Comparison with pulmonary function testing and other clinical measures

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krefft SD, Strand M, Smith J, Stroup C, Meehan R, Rose C. Utility of Lung Clearance Index Testing as a Noninvasive Marker of Deployment-related Lung Disease. J Occup Environ Med. 2017 Aug;59(8):707-711. doi: 10.1097/JOM.0000000000001058. PMID 28665837
- [Background] Zell-Baran LM, Krefft SD, Moore CM, Wolff J, Meehan R, Rose CS. Multiple breath washout test data for healthy controls. Data Brief. 2020 Dec 10;34:106641. doi: 10.1016/j.dib.2020.106641. eCollection 2021 Feb. PMID 33365370